CLINICAL TRIAL: NCT04256421
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of Atezolizumab Plus Carboplatin and Etoposide With or Without Tiragolumab (Anti-Tigit Antibody) in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of Atezolizumab Plus Carboplatin and Etoposide With or Without Tiragolumab in Patients With Untreated Extensive-Stage Small Cell Lung Cancer
Acronym: SKYSCRAPER-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GO41767; 2019-003301-97 (EudraCT Number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Tiragolumab; atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Atezolizumab + CE (Active Comparator): Participants will receive atezolizumab on Day 1 of each 21-day cycle followed by placebo on Day 1 of each 21-day cycle. Carboplatin will be administered followed by etoposide on Day 1 for 4 cycles. Participants will also receive etoposide on Days 2 and 3.
  Interventions: Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide; Drug: Placebo
- Tiragolumab + Atezolizumab + CE (Experimental): Participants will receive atezolizumab on Day 1 of each 21-day cycle followed by tiragolumab on Day 1 of each 21-day cycle. Carboplatin will be administered followed by etoposide on Day 1 for 4 cycles. Participants will also receive etoposide on Days 2 and 3.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Tiragolumab — Tiragolumab 600 milligrams (mg) administered by IV infusion on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A
  Arms: Tiragolumab + Atezolizumab + CE
Drug: Atezolizumab — Atezolizumab 1200 mg administered by IV infusion on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
Drug: Carboplatin — Carboplatin was administered by IV infusion on Day 1 of each 21-day cycle for 4 cycles.
Drug: Etoposide — Etoposide 100 mg/m^2 administered by IV infusion on Days 1, 2 and 3 of each 21-day cycle for 4 cycles.
Drug: Placebo — Placebo administered by IV infusion on Day 1 of each 21-day cycle.
  Arms: Placebo + Atezolizumab + CE

SUMMARY:
This study will evaluate the efficacy of tiragolumab plus atezolizumab and carboplatin and etoposide (CE) compared with placebo plus atezolizumab and CE in participants with chemotherapy-naive extensive-stage small cell lung cancer (ES-SCLC). Eligible participants will be stratified by Eastern Cooperative Oncology Group (ECOG) Performance Status (0 vs. 1), LDH (</= upper limit of normal [ULN] vs. > ULN), and presence or history of brain metastasis (yes vs. no) and randomly assigned in a 1:1 ratio to receive one of the following treatment regimens during induction phase:

* Arm A: Tiragolumab plus atezolizumab plus CE
* Arm B: Placebo plus atezolizumab plus CE

Following the induction phase, participants will continue maintenance therapy with either atezolizumab plus tiragolumab (Arm A) or atezolizumab plus placebo (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC)
* No prior systemic treatment for ES-SCLC
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
* Adequate hematologic and end-organ function
* Treatment-free for at least 6 months since last chemo/radiotherapy, among those treated (with curative intent) with prior chemo/radiotherapy for limited-stage SCLC

Exclusion Criteria:

* Symptomatic or actively progressing central nervous system (CNS) metastases
* Malignancies other than small cell lung cancer (SCLC) within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Positive test result for human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C
* Severe infection at the time of randomization
* Treatment with any other investigational agent within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-cytotoxic T lymphocyte-associated protein 4 (anti-CTLA-4), anti-TIGIT, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug elimination half-lives prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (121):
- United States (18):
  - Rocky Mountain Cancer Centers - Lone Tree, Lone Tree, Colorado
  - MedStar Georgetown University Hospital (Lombardi Comprehensive Cancer Center), Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - SCRI Florida Cancer Specialists North, Sarasota, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Illinois Cancer Care, Peoria, Illinois
  - New England Cancer Specialists, Scarborough, Maine
  - Weinberg Cancer Institution at Franklin Square, Baltimore, Maryland
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Broome Oncology - Binghamton, Binghamton, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute / Tennessee Oncology, Chattanooga, Tennessee
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Texas Oncology Cancer Center, Austin, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
- Austria (3):
  - Tiroler Landeskrankenanstalten Ges.M.B.H., Innsbruck
  - Klinik Penzing, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
- Belgium (4):
  - AZ St Maarten Campus Leopoldstr, Mechelen
  - Clinique Ste-Elisabeth, Namur
  - AZ Delta (Campus Rumbeke), Roeselare
  - Vitaz, Sint-Niklaas
- Brazil (6):
  - Oncocentro Serviços Médicos e Hospitalares Ltda, Fortaleza, Ceará
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital de Clínicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Clínica de Oncologia Reichow, Blumenau, Santa Catarina
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc
  - Vitkovicka Nemocnice Bma, A.S., Ostrava
  - Thomayerova nemocnice, Praha 4 - Krc
- Germany (6):
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - LungenClinic Großhansdorf GmbH, Großhansdorf
  - Asklepios Klinik Harburg, Hamburg
  - Fachklinik für Lungenerkrankungen, Immenhausen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Asklepios Klinik Gauting, München-Gauting
- Greece (4):
  - General Hospital "G.Papanikolaou", Asvestochóri
  - Uoa Sotiria Hospital, Athens
  - Metropolitan General Hospital, Cholargós
  - Univ General Hosp Heraklion, Heraklion
- Hungary (3):
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rend.Int., Szolnok
  - Tudogyogyintezet Torokbalint, Törökbálint
- Italy (7):
  - Irccs Ist. Tumori Giovanni Paolo Ii, Bari, Apulia
  - AORN Ospedali dei Colli Ospedale Monaldi, Napoli, Campania
  - AUSL della Romagna, Ravenna, Emilia-Romagna
  - IRCCS Istituto Clinico Humanitas, Rozzano, Lombardy
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Azienda Ospedaliero-Universitaria ?PoliclinicoVittorio Emanuele?- P.O. G. Rodolico, Catania, Sicily
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Japan (11):
  - National Cancer Center Hospital East, Chiba
  - Kyushu University Hospital, Fukuoka
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osaka
  - NHO Kinki-Chuo Chest Medical Center, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Erasmus MC, Rotterdam
- Auckland City Hospital, Auckland, New Zealand
- Poland (7):
  - Szpital Specjalistyczny Podkarpacki O?rodek Onkologiczny, Brzozów
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Krakowski Szpital Specjalistyczny im sw.Jana Pawla II, Krakow
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii w Poznaniu, Poznan
  - Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad, Warsaw
- Russia (3):
  - Principal Military Clinical Hospital n.a. N.N. Burdenko, Moscow, Moscow Oblast
  - Blokhin Cancer Research Center, Moscow, Moscow Oblast
  - Scientific Research Institute n.a. N.N. Petrov, Saint Petersburg, Sankt-Peterburg
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center ''Bezanijska Kosa'', Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (10):
  - Chungbuk National University Hospital, Cheongju-si
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Samsung Changwon Hospital, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (8):
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Switzerland (2):
  - CHUV, Lausanne
  - UniversitätsSpital Zürich, Zurich
- Taiwan (4):
  - National Cheng-Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Medical Foundation, Linkou Branch, Taoyuan District
  - National Taiwan University Hospital, Zhongzheng Dist.
- Turkey (Türkiye) (6):
  - Adana Baskent University Hospital, Adana
  - Ankara University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Istanbul University Cerrahpa?a-Cerrahpa?a Medical Faculty, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - ?zmir Medical Park, Izm?r
- United Kingdom (4):
  - NHS Lothian - Western General Hospital, Edinburgh
  - Guys and St Thomas Hospital, London
  - Christie Foundation Trust, Manchester
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Rudin CM, Liu SV, Soo RA, Lu S, Hong MH, Lee JS, Bryl M, Dumoulin DW, Rittmeyer A, Chiu CH, Ozyilkan O, Johnson M, Navarro A, Novello S, Ozawa Y, Tam SH, Patil NS, Wen X, Huang M, Hoang T, Meng R, Reck M. SKYSCRAPER-02: Tiragolumab in Combination With Atezolizumab Plus Chemotherapy in Untreated Extensive-Stage Small-Cell Lung Cancer. J Clin Oncol. 2024 Jan 20;42(3):324-335. doi: 10.1200/JCO.23.01363. Epub 2023 Nov 17. PMID 37976444

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 490 participants with extensive stage small cell lung cancer (SCLC) took part at 139 centers across 23 countries.
Pre-assignment Details: Participants were randomized to receive Placebo + Atezolizumab (P+A) or Tiragolumab + Atezolizumab (T+A) with carboplatin & etoposide as induction treatment followed by either P+A or T+A as maintenance treatment. 1 participant from P+A arm and 4 from T+A arm were randomized but not treated. Results from primary analysis are reported here. Final results of the study will be made public 1 year after study completion.
Groups:
- Placebo + Atezolizumab: During induction treatment participants received atezolizumab, 1200 milligram (mg) followed by placebo and carboplatin, as intravenous (IV) infusion, to achieve an initial target area under the concentration-time curve (AUC) of 5 milligram/milliliter/minute (mg/mL/min) on Day 1 of each 21-day cycle for 4 cycles. Etoposide 100 milligram per square meter (mg/m^2) was also administered as IV infusion on Days 1, 2 and 3 of each 21-day cycle for 4 cycles. Participants then received maintenance treatment with atezolizumab+ placebo on Day 1 of each 21-day cycle at the same dose as during induction treatment until disease progression or loss of clinical benefit.
- Tiragolumab + Atezolizumab: During induction treatment participants received atezolizumab, 1200 mg followed by tiragolumab, 600mg and carboplatin, as IV infusion, to achieve an initial target AUC of 5 mg/mL/min on Day 1 of each 21-day cycle for 4 cycles. Etoposide 100 mg/m^2 was also administered as IV infusion on Days 1, 2 and 3 of each 21-day cycle for 4 cycles. Participants then received maintenance treatment with atezolizumab+ tiragolumab on Day 1 of each 21-day cycle at the same dose as during induction treatment until disease progression or loss of clinical benefit.
Period: Overall Study
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Started | 247 | 243
Safety-evaluable Set (Safety-evaluable set included all randomized participants who received at least one dose of study treatment.) | 246 (1 participant from P+A arm was randomized but not treated.) | 239 (4 participants from T+A arm were randomized but not treated.)
Completed | 0 | 0
Not Completed | 247 | 243
Not completed — Death | 171 | 180
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Ongoing in Study | 66 | 52

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All randomized participants, whether or not the participant received the assigned treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab | Total
Number analyzed (Participants) | 247 | 243 | 490
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (7.9) | 64.5 (8.2) | 64.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 81 | 164
  Male | 164 | 162 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 10 | 17
  Not Hispanic or Latino | 229 | 224 | 453
  Unknown or Not Reported | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 67 | 63 | 130
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 2 | 1 | 3
  White | 174 | 173 | 347
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Investigator-Assessed Progression Free Survival (PFS) in the Primary Analysis Set (PAS)
Description: PFS was defined as the time from randomization to the first documented disease progression (PD) as determined by the investigator with the use of Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurred first. PD: at least a 20% increase in the sum of diameters (SOD) of target lesions, taking as reference the smallest SOD on study (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 24 months)
Population: Primary analysis set (PAS): All randomized participants without presence or history of brain metastases at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 201 | 196
months | 5.55 [5.36 to 5.85] | 5.36 [4.67 to 5.52]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> upper limit of normal [ULN] vs. </= ULN) and Eastern Cooperative Oncology Group (ECOG; 0 vs. 1); Test type: Superiority; p = 0.3504, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.89 to 1.38]

2. Primary Outcome: Overall Survival (OS) in the PAS
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause (up to approximately 24 months)
Population: PAS: All randomized participants without presence or history of brain metastases at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 201 | 196
months | 13.14 [12.16 to 15.11] | 13.11 [10.84 to 14.39]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.2859, Log Rank; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.90 to 1.44]

3. Secondary Outcome: PFS in the FAS
Description: PFS was defined as the time from randomization to the first documented PD as determined by the investigator with the use of RECIST v1.1 or death from any cause, whichever occurred first. PD: at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on study (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of >/= 5 mm.
Time Frame: as for outcome 1
Population: FAS: All randomized participants, whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 247 | 243
months | 5.42 [4.47 to 5.65] | 5.06 [4.40 to 5.42]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.4440, Log Rank; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.89 to 1.31]

4. Secondary Outcome: OS in the FAS
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause (up to approximately 24 months)
Population: FAS: All randomized participants, whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 247 | 243
months | 12.91 [11.99 to 14.52] | 12.75 [10.84 to 14.29]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.4205, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.88 to 1.35]

5. Secondary Outcome: Investigator-Assessed Confirmed Objective Response Rate (ORR) in the PAS
Description: ORR was defined as the percentage of participants with a complete response (CR) or a partial response (PR) as determined by the investigator with the use of RECIST v1.1. CR was defined as disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR.
Time Frame: From randomization up to approximately 24 months
Population: PAS: All randomized participants without presence or history of brain metastases at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 201 | 196
percentage of participants | 66.7 [59.64 to 73.05] | 73.5 [66.61 to 79.39]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.1418, Cochran-Mantel-Haenszel; Difference in Overall Response Rates = 6.80, 95% CI 2-sided [-2.57 to 15.99]

6. Secondary Outcome: Investigator-Assessed Confirmed ORR in the FAS
Description: ORR was defined as the percentage of participants with CR or PR as determined by the investigator with the use of RECIST v1.1. CR was defined as disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR.
Time Frame: From randomization up to approximately 24 months
Population: FAS: All randomized participants, whether or not the participant received the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 247 | 243
percentage of participants | 65.6 [59.26 to 71.42] | 70.8 [64.56 to 76.33]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.2191, Cochran-Mantel-Haenszel; Difference in Overall Response Rates = 5.19, 95% CI 2-sided [-3.33 to 13.61]

7. Secondary Outcome: Investigator-Assessed Duration of Response (DOR) in the PAS
Description: DOR was defined as the time from the first occurrence of a documented objective response (OR) to PD or death from any cause, whichever occurred first, as determined by the investigator with the use of RECIST v1.1. CR: was defined as disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to < 10 mm PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD= at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on study (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of >/= 5 mm.
Time Frame: From the first occurrence of a documented confirmed objective response to disease progression or death from any cause, whichever occurs first (up to approximately 24 months)
Population: PAS: All randomized participants without presence or history of brain metastases at baseline. DOR was analyzed in confirmed responders by investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 134 | 144
months | 5.59 [4.57 to 6.93] | 4.19 [4.14 to 4.60]

8. Secondary Outcome: Investigator-Assessed DOR in the FAS
Description: DOR was defined as the time from the first occurrence of a documented OR to PD or death from any cause, whichever occurred first, as determined by the investigator with the use of RECIST v1.1. CR: was defined as disappearance of all target lesions or any pathological lymph nodes must have reduction in short axis to < 10 mm PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD= at least a 20% increase in the SOD of target lesions, taking as reference the smallest SOD on study (including baseline). In addition to the relative increase of 20%, the SOD must also demonstrate an absolute increase of >/= 5 mm.
Time Frame: as for outcome 7
Population: FAS: All randomized participants, whether or not the participant received the assigned treatment. DOR was analyzed in confirmed responders by investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 162 | 172
months | 5.11 [4.37 to 5.75] | 4.17 [4.07 to 4.37]

9. Secondary Outcome: Investigator-Assessed PFS Rates at 6 Months and 12 Months in the PAS
Description: PFS rate at 6 months and 12 months was defined as the percentage of participants who were event free at these specific time points. Percentages have been rounded off to the nearest decimal point. A point estimate of the event-free rate is a single, numerical value used to approximate the true event-free rate of the entire population at a specific point in time. This value is calculated from ordered data (Event, Censoring) of each patient, using the Kaplan-Meier method, and accounts for censored observations( so Event free rates may not directly be calculated based only on patients remaining at risk).
Time Frame: Month 6, Month 12
Population: PAS: All randomized participants without presence or history of brain metastases at baseline. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 84 | 67
percentage of participants
  Month 6 | 42.42 [35.54 to 49.31] | 35.15 [28.41 to 41.90]
  Month 12: number analyzed (Participants) | 26 | 17
  Month 12 | 17.29 [11.90 to 22.69] | 14.21 [9.06 to 19.35]

10. Secondary Outcome: Investigator-Assessed PFS Rates at 6 Months and 12 Months in the FAS
Description: as for outcome 9
Time Frame: Month 6, Month 12
Population: FAS: All randomized participants, whether or not the participant received the assigned treatment. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 92 | 74
percentage of participants
  Month 6 | 37.95 [31.85 to 44.05] | 31.30 [25.41 to 37.19]
  Month 12: number analyzed (Participants) | 26 | 18
  Month 12 | 14.07 [9.59 to 18.55] | 12.33 [7.90 to 16.75]

11. Secondary Outcome: Overall Survival Rates at 12 Months and 24 Months in the PAS
Description: Overall survival rate at 12 months and 24 months was defined as the percentage of participants who were alive at these specific time points. Percentages have been rounded off to the nearest decimal point. A point estimate of the event-free rate is a single, numerical value used to approximate the true event-free rate of the entire population at a specific point in time. This value is calculated from ordered data (Event, Censoring) of each patient, using the Kaplan-Meier method, and accounts for censored observations( so Event free rates may not directly be calculated based only on patients remaining at risk).
Time Frame: Month 12, Month 24
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 112 | 103
percentage of participants
  Month 12 | 57.74 [50.82 to 64.66] | 54.00 [46.97 to 61.03]
  Month 24: number analyzed (Participants) | 12 | 10
  Month 24 | 27.68 [20.43 to 34.94] | 19.56 [13.16 to 25.96]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Month 12; Test type: Superiority; p = 0.4580, Z-test; Difference in Event Free Rate = -3.74, 95% CI 2-sided [-13.60 to 6.13]
Statistical Analysis 2: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Month 24; Test type: Superiority; p = 0.0999, Z-test; Difference in Event Free Rate = -8.12, 95% CI 2-sided [-17.80 to 1.55]

12. Secondary Outcome: Overall Survival Rates at 12 Months and 24 Months in the FAS
Description: as for outcome 11
Time Frame: Month 12, Month 24
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 133 | 125
percentage of participants
  Month 12 | 55.84 [49.58 to 62.10] | 52.82 [46.49 to 59.15]
  Month 24: number analyzed (Participants) | 12 | 10
  Month 24 | 25.82 [19.19 to 32.46] | 20.53 [14.54 to 26.52]
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Month 12; Test type: Superiority; p = 0.5059, Z-test; Difference in Event Free Rate = -3.02, 95% CI 2-sided [-11.92 to 5.88]
Statistical Analysis 2: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Month 24; Test type: Superiority; p = 0.2458, Z-test; Difference in Event Free Rate = -5.29, 95% CI 2-sided [-14.23 to 3.65]

13. Secondary Outcome: Time to Confirmed Deterioration (TTCD) of European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core (QLQ-C30) Physical Functioning in the PAS
Description: TTCD was the time from randomization until the first confirmed clinically meaningful deterioration in physical functioning. TTCD was determined based on patient-reported physical functioning (items 1-5) as collected and measured by the EORTC QLQ-C30. The PF is measured on 4-point scale (1='Not at all' to 4='Very much'). A high score for the physical function subscale represented a high/healthy level of functioning. The scale was linearly transformed so that each score ranged from 0 to 100. A score change of at least 10-point in physical functioning subscale score was perceived by participants as clinically meaningful. Confirmed clinically meaningful deterioration was defined as a clinically meaningful decrease from baseline that was held for at least two consecutive assessments or an initial clinically meaningful decrease from baseline followed by death from any cause within 3 weeks.
Time Frame: From randomization until the first confirmed clinically meaningful deterioration up to approximately 24 months
Population: PAS: All randomized participants without presence or history of brain metastases at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 201 | 196
months | 19.35 [19.35 to NA] — NA = not estimable due to an insufficient number of events | 15.67 [12.81 to NA] — NA = not estimable due to an insufficient number of events
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.9819, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.68 to 1.48]

14. Secondary Outcome: TTCD of EORTC QLQ-C30 Physical Functioning in the FAS
Description: as for outcome 13
Time Frame: From randomization until the first confirmed clinically meaningful deterioration up to approximately 24 months
Population: FAS: All randomized participants, whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 247 | 243
months | 19.35 [12.42 to NA] — NA = not estimable due to an insufficient number of events | 15.67 [11.83 to NA] — NA = not estimable due to an insufficient number of events
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.5122, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.81 to 1.55]

15. Secondary Outcome: TTCD of EORTC QLQ-C30 Global Health Status (GHS)/Quality of Life (QoL) in the PAS
Description: TTCD was the time from randomization until the first confirmed clinically meaningful deterioration in patient-reported global health status (GHS)/ quality of life (QoL). TTCD was determined based on patient-reported GHS/QoL (items 29-30) as collected and measured by the EORTC QLQ-C30. HS/QoL items are scored on a 7-point scale that ranges from "very poor" to "excellent". A high score for the GHS/QoL subscale represented a high health related quality of life. The scale was linearly transformed so that each score ranged from 0 to 100. A score change of at least 10-point in GHS/QoL subscale score was perceived by participants as clinically meaningful. Confirmed clinically meaningful deterioration was defined as a clinically meaningful decrease from baseline that was held for at least two consecutive assessments or an initial clinically meaningful decrease from baseline followed by death from any cause within 3 weeks.
Time Frame: From randomization until the first confirmed clinically meaningful deterioration up to approximately 24 months
Population: PAS: All randomized participants without presence or history of brain metastases at baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 201 | 196
months | NA [NA to NA] — NA = not estimable due to an insufficient number of events | NA [14.55 to NA] — NA = not estimable due to an insufficient number of events
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.3614, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.81 to 1.79]

16. Secondary Outcome: TTCD of EORTC QLQ-C30 GHS/QoL in the FAS
Description: TTCD was the time from randomization until the first confirmed clinically meaningful deterioration in patient-reported global health status (GHS)/ quality of life (QoL). TTCD was determined based on patient-reported GHS/QoL (items 29-30) as collected and measured by the EORTC QLQ-C30. HS/ QoL items are scored on a 7-point scale that ranges from "very poor" to "excellent". A high score for the GHS/QoL subscale represented a high health related quality of life. The scale was linearly transformed so that each score ranged from 0 to 100. A score change of at least 10-point in GHS/QoL subscale score was perceived by participants as clinically meaningful. Confirmed clinically meaningful deterioration was defined as a clinically meaningful decrease from baseline that was held for at least two consecutive assessments or an initial clinically meaningful decrease from baseline followed by death from any cause within 3 weeks.
Time Frame: From randomization until the first confirmed clinically meaningful deterioration up to 24 months
Population: FAS: All randomized participants, whether or not the participant received the assigned treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 247 | 243
months | NA [NA to NA] — NA = not estimable due to an insufficient number of participants with events | NA [14.55 to NA] — NA = not estimable due to an insufficient number of participants with events
Statistical Analysis 1: Comparison: Placebo + Atezolizumab vs Tiragolumab + Atezolizumab; Stratification factors were LDH (> ULN vs. </= ULN) and ECOG (0 vs. 1); Test type: Superiority; p = 0.1681, Log Rank; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.90 to 1.84]

17. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to 65 months
Reporting Status: Not Posted, anticipated posting 2026-07

18. Secondary Outcome: Minimum Serum Concentration (Cmin) of Tiragolumab
Time Frame: At the end of each cycle (each cycle is 21 days) of Cycles 1, 2, 3, 7, 11 and 15 (approximately 11 months)
Population: PK-evaluable set: All participants who received at least one dose of study treatment and who had at least one post-baseline PK sample available. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 218
microgram/milliliter (mcg/mL)
  Cycle 1 | 29.5 (49.2)
  Cycle 2: number analyzed (Participants) | 213
  Cycle 2 | 46.5 (47.5)
  Cycle 3: number analyzed (Participants) | 201
  Cycle 3 | 56.3 (83.5)
  Cycle 7: number analyzed (Participants) | 111
  Cycle 7 | 76.3 (48.2)
  Cycle 11: number analyzed (Participants) | 45
  Cycle 11 | 78.8 (246)
  Cycle 15: number analyzed (Participants) | 17
  Cycle 15 | 96.4 (43.8)

19. Secondary Outcome: Cmin of Atezolizumab
Time Frame: At the end of each cycle (each cycle is 21 days) of Cycles 1, 2, 3, 7, 11 and 15 (approximately 11 months)
Population: PK-evaluable set: All participants who received at least one dose of study treatment and who had at least one post-baseline PK sample available. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 226 | 217
mcg/mL
  Cycle 1 | 75.0 (63.2) | 75.4 (70.8)
  Cycle 2: number analyzed (Participants) | 221 | 213
  Cycle 2 | 121 (55.8) | 125 (38.4)
  Cycle 3: number analyzed (Participants) | 200 | 198
  Cycle 3 | 144 (49.8) | 155 (81.5)
  Cycle 7: number analyzed (Participants) | 115 | 110
  Cycle 7 | 205 (45.3) | 198 (46.4)
  Cycle 11: number analyzed (Participants) | 52 | 45
  Cycle 11 | 226 (37.3) | 244 (37)
  Cycle 15: number analyzed (Participants) | 26 | 17
  Cycle 15 | 198 (75.5) | 253 (36.6)

20. Secondary Outcome: Maximum Serum Concentration (Cmax) of Tiragolumab
Time Frame: Predose and 30 minutes post end of infusion (EOI) on Day 1 of Cycle 1 (each cycle is 21 days)
Population: PK-evaluable set: All participants who received at least one dose of study treatment and who had at least one post-baseline PK sample available. Overall number of participants analyzed is the number of participants with data available for analyses
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 213
mcg/mL | 188 (24.2)

21. Secondary Outcome: Cmax of Atezolizumab
Time Frame: Predose and 30 minutes post EOI on Day 1 of Cycle 1 (each cycle is 21 days)
Population: PK-evaluable set: All participants who received at least one dose of study treatment and who had at least one post-baseline PK sample available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 233 | 224
mcg/mL | 398 (28.2) | 405 (23.0)

22. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Tiragolumab
Description: Reported here is the number of participants who had a positive ADA assay result at baseline and the number of participants positive for treatment emergent ADAs. The participants positive for treatment emergent ADAs include treatment-induced and treatment-enhanced ADA positive participants. Treatment-induced ADAs are participants with negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADAs are participants with a positive ADA result at baseline who had one or more post-baseline titer results that were at least 0.60 t.u. greater than the baseline titer result. The total number of participants who developed ADAs to tiragolumab was determined by summing the ADA-positive participants across all timepoints.
Time Frame: Predose on Day 1 of Cycles 1 (each cycle is 21 days), 2, 3, 4, 8,12 and 16 and at treatment discontinuation (TD) visit (up to 24 months)
Population: Tiragolumab ADA-evaluable set: All participants who received at least one dose of tiragolumab treatment and with an ADA assay result from at least one sample result. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 235
Participants
  Participants with Positive Sample at Baseline | 2
  Participants positive for Treatment Emergent ADAs: number analyzed (Participants) | 229
  Participants positive for Treatment Emergent ADAs | 3
  Treatment-induced ADAs: number analyzed (Participants) | 229
  Treatment-induced ADAs | 3
  Treatment-enhanced ADAs: number analyzed (Participants) | 229
  Treatment-enhanced ADAs | 0

23. Secondary Outcome: Number of Participants With ADAs to Atezolizumab
Description: Reported here is the number of participants who had a positive ADA assay result at baseline and the number of participants positive for treatment emergent ADAs. The number of participants positive for treatment emergent ADAs includes treatment-induced and treatment-enhanced ADA positive participants. Treatment-induced ADAs are participants with negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADAs are participants with a positive ADA result at baseline who had one or more post-baseline titer results that were at least 0.60 t.u. greater than the baseline titer result. The total number of participants who developed ADAs to atezolizumab was determined by summing the ADA-positive participants across all timepoints.
Time Frame: Predose on Day 1 of Cycles 1 (each cycle is 21 days), 2, 3, 4, 8,12 and 16 and at TD visit (up to 24 months)
Population: Atezolizumab ADA-evaluable set: All participants who received at least one dose of atezolizumab treatment and with an ADA assay result from at least one sample result. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
Number analyzed (Participants) | 244 | 236
Participants
  Participants with Positive Sample at Baseline | 2 | 1
  Participants positive for Treatment Emergent ADAs: number analyzed (Participants) | 238 | 228
  Participants positive for Treatment Emergent ADAs | 48 | 22
  Treatment-induced ADAs: number analyzed (Participants) | 238 | 228
  Treatment-induced ADAs | 48 | 22
  Treatment-enhanced ADAs: number analyzed (Participants) | 238 | 228
  Treatment-enhanced ADAs | 0 | 0

24. Secondary Outcome: Change From Baseline in EuroQol 5-Dimension, 5-Level (EQ-5D-5L) Index-based and Visual Analog Scale Scores
Description: The EQ-5D-5L is a validated self-report health status questionnaire that was used to calculate a health status utility score for use in health economic analyses. There were two components to the EQ-5D-5L: a five-item health state profile that assessed mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, as well as a visual analog scale (VAS) that measured health state. The EQ VAS records the participant's self-rated health on a vertical visual analogue scale ranging from 0 to 100 A single composite score was calculated based on the responses as an indicator of the participant's health status. The scale ranges 0-100, 0=worst health and 100=best health.
Time Frame: From baseline up to 65 months
Reporting Status: Not Posted, anticipated posting 2026-07

ADVERSE EVENTS:
Time Frame: Up to approximately 24 months
Description: All-cause mortality- FAS: All randomized participants, whether or not the participant received the assigned treatment. SAE & other AEs: Safety-evaluable set included all randomized participants who received at least one dose of study treatment. All-cause mortality is reported for all randomized participants, whether or not the participant received the assigned treatment.
Arm/Group | Placebo + Atezolizumab | Tiragolumab + Atezolizumab
All-Cause Mortality (participants affected / at risk) | 171/247 | 180/243
Serious Adverse Events (participants affected / at risk) | 104/246 | 108/239
Other Adverse Events (participants affected / at risk) | 233/246 | 228/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Atezolizumab (N=246) | Tiragolumab + Atezolizumab (N=239)
Anaemia (Blood and lymphatic system disorders) | 8 (10) | 9 (10)
Bicytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 14 (15) | 16 (17)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (4) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 1 (4)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 9 (9) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (2) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 12 (15) | 7 (8)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (4) | 4 (4)
Platelet count decreased (Investigations) | 2 (2) | 3 (3)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 9 (17)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2) | 3 (3)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Limbic encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1)
Neuromyotonia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Mental disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Atezolizumab (N=246) | Tiragolumab + Atezolizumab (N=239)
Anaemia (Blood and lymphatic system disorders) | 97 (127) | 86 (106)
Leukopenia (Blood and lymphatic system disorders) | 13 (21) | 13 (17)
Neutropenia (Blood and lymphatic system disorders) | 72 (136) | 63 (91)
Thrombocytopenia (Blood and lymphatic system disorders) | 31 (53) | 29 (46)
Hyperthyroidism (Endocrine disorders) | 17 (19) | 16 (16)
Hypothyroidism (Endocrine disorders) | 21 (27) | 26 (26)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 12 (19)
Constipation (Gastrointestinal disorders) | 61 (67) | 58 (67)
Diarrhoea (Gastrointestinal disorders) | 37 (46) | 20 (24)
Nausea (Gastrointestinal disorders) | 61 (73) | 59 (66)
Vomiting (Gastrointestinal disorders) | 26 (36) | 21 (27)
Asthenia (General disorders) | 34 (46) | 23 (29)
Chest pain (General disorders) | 13 (14) | 9 (9)
Fatigue (General disorders) | 48 (61) | 59 (70)
Oedema peripheral (General disorders) | 11 (14) | 13 (16)
Pyrexia (General disorders) | 25 (26) | 17 (17)
COVID-19 (Infections and infestations) | 17 (17) | 13 (13)
Infusion related reaction (Injury, poisoning and procedural complications) | 17 (23) | 32 (39)
Alanine aminotransferase increased (Investigations) | 15 (20) | 17 (21)
Aspartate aminotransferase increased (Investigations) | 13 (16) | 14 (18)
Neutrophil count decreased (Investigations) | 55 (99) | 50 (89)
Platelet count decreased (Investigations) | 24 (32) | 27 (41)
Weight decreased (Investigations) | 15 (17) | 11 (11)
White blood cell count decreased (Investigations) | 26 (47) | 28 (50)
Decreased appetite (Metabolism and nutrition disorders) | 38 (50) | 58 (62)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (24) | 11 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 (24) | 14 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (17) | 20 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (27) | 20 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (19) | 17 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (17)
Dizziness (Nervous system disorders) | 22 (23) | 13 (15)
Headache (Nervous system disorders) | 17 (20) | 18 (20)
Insomnia (Psychiatric disorders) | 18 (19) | 29 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 18 (20)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (35) | 19 (20)
Alopecia (Skin and subcutaneous tissue disorders) | 67 (68) | 62 (62)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 12 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (34) | 66 (76)
Rash (Skin and subcutaneous tissue disorders) | 28 (33) | 36 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04256421/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT04256421/SAP_001.pdf